CLINICAL TRIAL: NCT05795283
Title: Potential Predictive Biological Markers of Major Depression Response to Citalopram Therapy in Patients With Anorexia Nervosa: a Single-center Study.
Brief Title: Potential Predictive Biological Markers of Major Depression Response to Citalopram Therapy in Anorexia Nervosa.
Acronym: ANCITA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 21C222
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Anorexia Nervosa
Keywords: Major depression; Citalopram; Biological markers
MeSH Terms: conditions — Anorexia Nervosa; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Citalopram i.v. and p.o: Both intravenous and oral administration of citalopram
  Interventions: Drug: Citalopram i.v. and p.o
- Group B: Citalopram p.o: Oral administration of citalopram
  Interventions: Drug: Citalopram p.o

INTERVENTIONS:
Drug: Citalopram i.v. and p.o — Citalopram:
  i.v.: 10 mg/die for day 1-7, 20 mg/die for day 8-14 p.o.: 20 mg/die for day 15-28
  Groups: Group A: Citalopram i.v. and p.o
Drug: Citalopram p.o — Citalopram:
  p.o: 10 mg/die for day 1-7, 20 mg/die for day 15-28
  Groups: Group B: Citalopram p.o

SUMMARY:
In patients suffering from anorexia nervosa associated with severe major depression, serotonin reuptake inhibitor drugs have shown little efficacy in significantly reducing depressive symptoms. A possible explanation for this poor efficacy could be that people with anorexia nervosa have a deficiency in amino acids such as tryptophan, which is necessary for the production of the neurotransmitter serotonin. Therefore, tryptophan supplementation has been suggested as a means of increasing the pharmacological response to serotonin reuptake inhibitor drugs in patients with anorexia nervosa. Furthermore, malnutrition present in patients suffering from anorexia nervosa is in some cases associated with problems of intestinal absorption of nutrients, with possible implications on the pharmacokinetics of the drugs administered, including selective serotonin reuptake inhibitors (SSRIs).

The present observational study aims to evaluate the correlations between the clinical response to Citalopram therapy (in different o.s. and i.v. formulations) and some nutritional, neurotransmitter and inflammatory biomarkers, in order to identify potential predictive markers of response to therapy for severe major depression in patients with anorexia nervosa.

The following parameters will be evaluated in patients enrolled in all 3 observation times described above:

* Plasma concentration of Citalopram
* Serum concentration of Serotonin
* Plasma concentration of dopamine
* Serum concentration of Tryptophan
* Serum concentration of BDNF
* Hamilton scale 17 items and other clinical scales (EDI-3, SCL-90, BUT).

ELIGIBILITY:
Inclusion Criteria:

* Anorexia nervosa
* Severe depression (Hamilton score 25 or higher)
* Written informed consent

Exclusion Criteria:

* Other psychiatric disorders
* Acute infectious diseases
* Chronic inflammatory diseases
* Disorders of central nervous system
* Pregnancy ore breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with anorexia nervosa and severe depression
Sampling Method: Non-Probability Sample
Enrollment: 123 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale | At baseline, 2 weeks and 4 weeks after treatment with citalopram
  17-item Hamilton Depression Rating Scale -
Change in plasma level of citalopram | At baseline, 2 weeks and 4 weeks after treatment with citalopram
  Plasma level of citalopram
Change in plasma level of dopamine | At baseline, 2 weeks and 4 weeks after treatment with citalopram
  Plasma level of dopamine
Change in serum level of serotonin | At baseline, 2 weeks and 4 weeks after treatment with citalopram
  Serum level of serotonin
Change in serum level of brain-derived neurotrophic factor | At baseline, 2 weeks and 4 weeks after treatment with citalopram
  Serum level of brain-derived neurotrophic factor
Change in serum level of tryptophan | At baseline, 2 weeks and 4 weeks after treatment with citalopram
  Serum level of tryptophan

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Oggebbio, Italy